CLINICAL TRIAL: NCT00711321
Title: Phase Ib Follow-up Study to Evaluate Long-term Safety and Tolerability of Immunization With AFFITOPE AD02 Applied During AFFiRiS 002
Brief Title: Long-term Safety and Tolerability of AFFITOPE AD02
Status: Completed | Type: Observational
Sponsor: Affiris AG (Industry)
Responsible Party: Affiris AG
Other Study IDs: Affiris 004; EudraCT 2008-002764-33
Record Dates: First submitted 2008-07-04; First posted 2008-07-08 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer; Morbus Alzheimer; Vaccine; Alzheimer Vaccine; A-beta immunotherapy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 2: AFFITOPE AD02 with adjuvant
- 1: AFFITOPE AD02 without adjuvant

SUMMARY:
The purpose of this study is to evaluate the long-term tolerability and -safety of AFFITOPE AD02 applied during AFFiRiS 002

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed and dated by patient and caregiver
* Patients having participated in AFF002 and having received at least 1 vaccination with AFFITOPE AD02
* Availability of a partner/caregiver knowing the patient and being able to accompany the patient to the visits

Exclusion Criteria:

* Patients having received no vaccination with AFFITOPE AD02
* History of questionable compliance to visit schedule, patients not expected to finish the clinical trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects having participated in AFFiRiS 002
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Long-term tolerability | 1 year

SECONDARY OUTCOMES:
Clinical and immunological efficacy (evaluated in an explorative manner only) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Margot Schmitz, MD Univ. D., Principal Investigator — Ordination Schmitz
Locations (1):
- Ordination Schmitz, Vienna, Austria